CLINICAL TRIAL: NCT05645445
Title: The Effect of Virtual Reality Application on Pain and Anxiety Level in Stone Crushing With Shock Waves: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Meral3
Record Dates: First submitted 2022-12-02; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Shockwave Lithotripsy; Pain; Anxiety; Virtual Reality; Nursing
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The routine ESWL procedure will be applied. Pre-procedural anxieties will be evaluated with the State-Trait Anxiety Inventory-State Anxiety Scale. After the ESWL procedure, their anxiety will be re-evaluated with the same scale, and their pain will also be evaluated with the Visual Analog Scale.
- virtual reality group (Experimental): The pre-procedure anxiety of the patients who will use virtual reality glasses during the ESWL process will be evaluated with the State-Trait Anxiety Inventory-State Anxiety Score. After the ESWL procedure, their anxiety will be re-evaluated with the same scale and in addition to the pain, the pain will be evaluated with the Visual Analog Scale.
  Interventions: Device: virtual reality

INTERVENTIONS:
Device: virtual reality — patients who include intervention gruop during the ESWL process, patients will be shown videos with virtual reality glasses, which include nature and landscapes, giving people a feeling of comfort and peace, and making them feel like they are inside.
  Arms: virtual reality group

SUMMARY:
This research was planned as a randomized controlled experimental study in order to evaluate the effect of virtual reality application on pain and anxiety caused by the procedure during stone crushing process (ESWL) with shock waves.

DETAILED DESCRIPTION:
Although urinary tract stones often remain asymptomatic at first, they can cause pain, hematuria, infection, decreased kidney function and kidney failure over time and can seriously affect the quality of life of people if not treated with appropriate methods.

Extracorporeal shockwave lithotripsy (ESWL) has been practiced as a treatment method to remove urolithiasis from the kidneys and ureters since the early 1980s.

The process is based on the principle that the sound waves obtained from a source other than the body are turned into shock waves and sent to the stone and the stone is broken down.

Relief of pain and anxiety during ESWL; In addition to maintaining patient comfort and satisfaction, it is extremely important to reduce the movement of the patient during the procedure and to facilitate the imaging and targeting of the stone.

Diverting attention is one of the most preferred methods to reduce the pain that occurs in patients while the diagnosis and treatment procedures are carried out. This method; It is a method that focuses the attention of patients on a different point and keeps the symptoms they experience under control and reduces them.

Strategies to divert attention include the application of virtual reality, which has been one of the methods that have attracted attention in recent years.

The individual focuses his attention on the image by moving away from real life with the glasses connected to the device worn on his head and the sounds coming from the headphones and feels as if he is in a different world thanks to these glasses.

In practice, it is aimed to reduce the patient's pain, discomfort and anxiety by drawing the patient's attention from pain and painful treatment procedures to a fun virtual environment.

ELIGIBILITY:
Inclusion Criteria:

* Applying to the stone crushing unit for the first time
* Body mass index below 30
* Those aged 18-65 who are literate and have no vision or hearing problems
* Have not taken any analgesics other than the analgesic routinely administered before the procedure

Exclusion Criteria:

* Untreated urinary tract infections
* Severe skeletal system malformations that prevent focusing on the stone
* Severe obesity
* Arterial aneurysm near the stone
* Patients with anatomical obstruction conditions in the distal part of the stone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
pain levels | one day
  pain measurement will be made by visual analog scale (VAS). The intensity will measure the area in which the individual mark between 0 (no pain) and 10 (worst pain i felt my life). The pain level will be asked one times before the shockwave process.
anxiety | one day
  Anxiety levels will be measure by the State-Trait Anxiety Inventory-State Anxiety (STAI-SA). The STAI scores were calculated based on the patients' answers. The overall score ranges from 20-80 and the higher the score indicates the higher the anxiety level. Patients with the STAI scores of 35 or lower were considered as having 'no anxiety' while patients with scores of 42 or higher were considered as 'severely anxious' as recommended by the practice guidelines. The survey will be used before and after shockwave for measure the anxiety levels in two groups.

CONTACTS AND LOCATIONS:
Overall Officials: meral Yıldırım Çetinkaya, PhD, Principal Investigator — Duzce University

IPD SHARING:
Plan to Share IPD: No